

#### STATISTICAL ANALYSIS PLAN FOR PROTOCOL AMP-518

Clinical Trials.gov Identifier: NCT05592418

**Sponsor:** 

AIM ImmunoTech Inc. 2117 SW Highway 484 Ocala, FL 34473, USA

Phone: Fax:

**Protocol Number:** AMP-518

Protocol Title: A Randomized, Double Blind, Placebo Controlled Study to

Evaluate the Efficacy and Safety of Ampligen® in Patients

with Post-COVID Conditions

**Protocol Version / Date:** Version 4.0/ Aug-23-2023

SAP Author: Amarex Clinical Research,

LLC

20201 Century Boulevard Germantown, MD 20874

USA

Telephone:

Facsimile:

**Plan Version:** SAP – Final Version 1.1

Plan Date: 6-Dec-2023

I

| <b>Protocol Number:</b> | AMP-518 |
|---|---|
| Protocol Version / Date: | Version 4.0/ Aug-23-2023 |
| Protocol Name: | A Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Ampligen® in Patients with Post-COVID Conditions |
| Sponsor: | AIM ImmunoTech Inc.<br>2117 SW Highway 484<br>Ocala, FL 34473, USA |
| Prepared by: | Amarex Clinical Research<br>20201 Century Boulevard<br>Germantown, Maryland 20874 |
| SAP Version: | SAP – Final Version 1.1 |
| SAP Date: | 6-Dec-2023 |
| I have read and approve the content: | e Statistical Analysis Plan specified above and agree on its |
| Statistician, Amarex Clinic | al Research Date |
| AIM ImmunoTech Inc. | Date |

#### TABLE OF CONTENTS

| Secti | on | | | Page |
|---|---|---|---|---|
| ABB | REVIAT | IONS, AC | CRONYMS, AND DEFINITIONS | 5 |
| 1. | | | ON | |
| 2. | PRO' | TOCOL D | DESIGN | 6 |
| | 2.1 | Design | Overview | 6 |
| | | 2.1.1 | Study Design | |
| | | 2.1.2 | Study Visits | |
| | 2.2 | | ent Groups | |
| | 2.3 | | mization and Stratification | |
| | 2.4 | | g | |
| | | 2.4.1<br>2.4.2 | Emergency Un-BlindingFinal Analysis | |
| | 2.5 | | ol Objective(s) | |
| | 2.6 | | y Assessments/ Outcome Measures | |
| | 2.0 | 2.6.1 | Primary Efficacy Outcome Measure | |
| | | 2.6.2 | Secondary Efficacy Outcome Measures | 12 |
| | | 2.6.3 | Exploratory Efficacy Outcome Measures | |
| | | 2.6.4 | Safety Outcome Measures | |
| 3. | | | E DETERMINATION, STATISTICAL POWER, AND SIGNIFIC | |
| 4. | INTE | RIM ANA | ALYSIS | 13 |
| 5. | PRIN | IARY HY | POTHESIS TO BE TESTED | 13 |
| 6. | ANA | LVSIS PO | PULATIONS | 13 |
| 0. | 711 171 | | | |
| 7. | DAT | A CONVE | ENTION AND RELATED DEFINITIONS | 4.4 |
| 7. | | | DEFINITION AND RELATED DEFINITIONS | |
| | 7.1<br>7.2 | | ate Data | |
| | – | | | |
| | 7.3 | 7.3.1 | ng of Missing Data | |
| | | 7.3.1 | Handling of Missing Data for Safety Evaluations | |
| | 7.4 | Multice | enter Clinical Trials | |
| | 7.5 | | le Comparisons and Multiplicity | |
| | 7.6 | _ | ates and Prognostic Factors | |
| | 7.7 | | ups | |
| | 7.8 | _ | rd Calculations | |
| | 7.0 | 7.8.1 | Body Mass Index (BMI) | |
| | | 7.8.2 | Change from baseline | 16 |
| | | 7.8.3 | Duration (days) of hospitalization during the treatment phase | 16 |
| 8. | STA | TISTICAL | METHODS | 17 |
| | 8.1 | Summa | arizing Disposition and Baseline Data | 17 |
| | | 8.1.1 | Subject Disposition and Withdrawals | 17 |
| | | 8.1.2 | Protocol Deviations | 17 |

| | | 8.1.3 | Demographics and Baseline Characteristics | 18 |
|-----|------|----------|---------------------------------------------|----|
| | | 8.1.4 | Medical History | |
| | | 8.1.5 | Prior and Concomitant Medications | 18 |
| | | 8.1.6 | Extent of Exposure and Treatment Compliance | 19 |
| | 8.2 | Analysi | is of Efficacy Data | 19 |
| | | 8.2.1 | Primary Outcome Measure and Estimand | |
| | | 8.2.2 | Secondary Outcome Measures | |
| | | 8.2.3 | Exploratory Outcome Measures | 23 |
| | 8.3 | Analysi | is of Safety Data | 24 |
| | | 8.3.1 | Adverse Events | 25 |
| | | 8.3.2 | Clinical Laboratory Evaluations | 25 |
| | | 8.3.3 | Vital Signs | |
| | | 8.3.4 | Electrocardiogram (ECGs) | 27 |
| | | 8.3.5 | Pulse Oxygen Saturation (SpO2) | 28 |
| | | 8.3.6 | Physical Examination | 28 |
| | | 8.3.7 | Urine Pregnancy Test | 28 |
| | | 0.2.0 | CARC C H 2 (COMP 10) O I'm' T | |
| | | 8.3.9 | SARS-CoV-2 (COVID-19) Qualitative Test | |
| | | 8.3.10 | COVID-19 History | |
| 9. | APPE | NDIX 1 | | 30 |
| 10. | APPE | NDIX 2 | | 36 |
| | 10.1 | Planned | d by-subject listings | 36 |
| | 10.2 | Plannec | d Summary Tables | 37 |
| 11. | APPE | NDIX 3 | | 38 |
| | 11.1 | PROM | IS FATIGUE SCORING TABLE | 38 |
| | 11.2 | PROM | IS COGNITIVE FUNCTION SCORING TABLE | 39 |
| | 11.3 | PROM | IS SLEEP DISTURBANCE SCORING TABLE | 40 |
| 12. | REFE | ERENCES | S | 41 |
| 13. | VERS | SION HIS | TORY | 42 |

#### ABBREVIATIONS, ACRONYMS, AND DEFINITIONS

**Abbreviation/Acronym Definition** 

ADSL Subject-Level Analysis Dataset

ALT Alanine Transaminase

Amarex Clinical Research, LLC.

ANC Absolute Neutrophil Count

ASA American Statistical Association
AST Aspartate Aminotransferase

BMI Body Mass Index

COVID Coronavirus Disease 2019

CRO Contract Research Organization

CSR Clinical Study Report

CTMS Clinical Trial Management System

ECG Electrocardiogram
EOT End of Treatment

FDA U.S. Food and Drug Administration

HCT Hematocrit

ICH International Conference on Harmonization

ITT Intention to Treat

IWRS Interactive Web Based Response System

IV Intravenous

LDH Lactate dehydrogenase

MoCA Montreal Cognitive Assessment

MCID Minimal Clinically Important Difference

PHQ Patient Health Questionnaire

RBC Red Blood Cells

SAE Serious Adverse Event

SARS Severe Acute Respiratory Syndrome

SAS Statistical Analysis System

SBQ-LC Symptom Burden Questionnaire for Long COVID

SLE Systemic Lupus Erythematosus

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

WBC White Blood Cells

#### 1. INTRODUCTION

This Statistical Analysis Plan describes the planned analyses and reporting for the clinical trial protocol AMP-518, conducted by AIM ImmunoTech Inc.. The reader of this Statistical Analysis Plan (SAP) is encouraged to review the complete protocol and amendments as this plan contains only a limited overview of protocol information. The main objectives of this plan are to provide details pertaining to statistical methodology, data conventions, and processes used for the analysis of data from this trial.

The format and content of this SAP are structured to provide sufficient detail to meet the requirements specified by the International Council on Harmonization (ICH) E9: Guidance on Statistical Principles in Clinical Trials. All work planned and presented in this Statistical Analysis Plan will follow the ethical guidelines published by the American Statistical Association (ASA).

The following documents were reviewed in preparation of this Statistical Analysis Plan:

- Protocol Version 4.0/ Aug-23-2023
- ASA Ethical Guidelines for Statistical Practice (2016)
- The Royal Statistical Society: Code of Conduct (2014)
- ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3, 1996)
- ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3(R1), 2013)
- ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9, 1998)
- ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9(R1), 2017)

#### 2. PROTOCOL DESIGN

#### 2.1 Design Overview

#### 2.1.1 Study Design

This is a Phase 2, two-arm, randomized, double blind, placebo controlled multicenter study to evaluate the efficacy and safety of Ampligen® in patients experiencing the Post-COVID Condition of fatigue. Patients will be randomized 1:1 to receive twice weekly IV infusions of Ampligen® or placebo.

Ampligen® and placebo will be administered via twice weekly infusions (Example:





# 2.1.1.3 Dosage Modification

### 2.1.2 Study Visits

#### 2.1.2.1 Study Schedule

The study will have three phases: Screening Phase, Treatment Phase, and Follow-Up Phase.

#### **Screening Phase (up to 1 week):**

All subjects will provide written informed consent and have a Screening visit (V1) within 7 days prior to first treatment visit (V2) to determine eligibility for subject participation.

All subjects who fail to meet eligibility criteria are considered screen failures and are exited from the study without further evaluation.

#### **Treatment Phase (12 weeks):**

Ampligen® and placebo will be administered via twice weekly infusions (Example: Monday/Thursday or Tuesday/Friday schedule) for 12 weeks.

#### Follow-Up Phase (2 weeks):

Two safety follow-up visits will be performed 3 to 4 days and 2 weeks after the End of Treatment (EOT) visit (V25).

#### 2.1.2.2 Unscheduled Visits

In the event that the subject will return to clinic at a time other than a regularly scheduled study visit, the visit will be regarded as an unscheduled visit. Assessments at unscheduled visits are at the discretion of the Investigator. All pertinent findings, including adverse events or changes in medications, will be noted in the eCRF.

# 2.2 Treatment Groups

| The following treatm | ent groups will be as | sessed in the study |
|----------------------|-----------------------|---------------------|
|----------------------|-----------------------|---------------------|

- Ampligen®
- Placebo (normal saline)

| A tota | al of 80 subjects (40 per | group) will be | e randomized in | n a 1:1 ratio | (Ampligen®: |
|---|---|---|---|---|---|
| placeb | 00). | | | | |
| 2.4 | Blinding | | | | |
| | s a double-blind study. The study is a double-blind study conduct | | | | sor/CRO staff |

#### 2.4.1 Emergency Un-Blinding

| Breaking the blind prematurely will be allowed only if the subject's well-being requires |
|---|
| knowledge of the subject's treatment allocation. Every attempt will be made to maintain |
| the blind throughout the study. |
| 2.4.2 Final Analysis |
| 2.4.2 Tiliai / tilaiy 515 |

# 2.5 Protocol Objective(s)

The purpose of this study is to assess the efficacy and safety of Ampligen® administered twice weekly by IV infusions in subjects experiencing the Post-COVID Condition of fatigue.

# 2.6 Efficacy Outcome Measures

## 2.6.1 Primary Efficacy Outcome Measure

• Change from baseline to week 13 in PROMIS® Fatigue Score (T-Score).

#### 2.6.2 Secondary Efficacy Outcome Measures

• Change from baseline to week 6 in PROMIS® Fatigue Score (T-Score).

Note: Additional PROMIS® Fatigue Score analysis (change from baseline) at week 6 and 13 will be performed excluding response to item, "How often did you have enough energy to exercise strenuously?"

- Change from baseline to week 6 and 13 in distance traveled during a 6-minute walk test.
- Proportion of subjects with minimal clinically important difference (MCID), defined as at least 54 m, in the Six-Minute Walk Test (6MWT) at the end of 12-week treatment phase.
- Change from baseline to week 6 and 13 in PROMIS® Cognitive Function Score (T-Score).
- Change from baseline to week 6 and 13 in PROMIS® Sleep Disturbance Score (T-Score).

#### 2.6.3 Exploratory Outcome Measures

• Changes from baseline in COVID-19-related symptoms using Symptom Burden Questionnaire for Long COVID (SBQ-LC) during the course of the treatment phase.

Note: A set of common COVID-19-related symptoms (see Symptom Burden Questionnaire for Long COVID (SBQ-LC)) will be evaluated at each scheduled study visit by the patient regardless of which symptoms a subject had at baseline, as new symptoms may appear following the baseline assessment.

- Change from baseline in cognitive function as measured by Montreal Cognitive Assessment (MoCA) at week 4, 8, and 13 during the treatment phase.
- Incidence of hospitalization during the treatment phase.
- Duration (days) of hospitalization during the treatment phase.
- Evaluation of lymphocyte profile by flow cytometry in patients with post-COVID-19 conditions.

• Identification and evaluation of plasma protein biomarkers in patients with post-COVID-19 conditions.

#### 2.6.4 Safety Outcome Measures

- Incidence of treatment-related adverse events.
- Incidence and severity of treatment-emergent adverse events (TEAEs).
- Incidence of serious adverse events (SAEs).
- Incidence of TEAEs and SAEs leading to discontinuation of study medication.
- Changes in blood chemistry, hematology, and coagulation results.
- Changes in vital signs including temperature, pulse, respiratory rate, systolic and diastolic blood pressure.
- Changes in physical examination results.
- Change in electrocardiogram (ECG) results.

# 3. SAMPLE SIZE DETERMINATION, STATISTICAL POWER, AND SIGNIFICANCE LEVEL

The sample size of 80 subjects will be used in this study. The sample size is based on clinical judgment. No statistical power calculation is used to establish the sample size for this proof-of-concept study.

#### 4. INTERIM ANALYSIS

There is no planned interim analysis for this early phase study.

#### 5. PRIMARY HYPOTHESIS TO BE TESTED

There is no formal hypothesis testing for this study as the study is a Phase II evaluation and is not intended to be hypothesis generating. The study is not powered to reliably yield statistically significant conclusions.

#### 6. ANALYSIS POPULATIONS



For all parameters, baseline will be defined as the last available value before the first randomized treatment.

# 7.2 Duplicate Data

#### 7.3 Handling of Missing Data

#### 7.3.1 Handling of Missing Data for Efficacy Evaluations

Every effort will be made to obtain required data at each scheduled evaluation from all subjects who have been randomized to minimize missing data.

#### 7.3.2 Handling of Missing Data for Safety Evaluations

The below imputation rules will be followed for imputation of missing dates:





#### 7.4 Multicenter Clinical Trials

This is a multi-center clinical trial.

# 7.5 Multiple Comparisons and Multiplicity

There will be no adjustment for multiple testing or multiplicity for this phase II trial. For all effectiveness endpoints, inference will be based on type I error rate of 0.05.

# 7.6 Covariates and Prognostic Factors

In the efficacy analysis, the stratification factors and baseline values will be used as

covariates in the analysis of all the primary, secondary, and additional efficacy endpoints.

#### 7.7 Subgroups



#### 7.8 Standard Calculations

#### 7.8.1 Body Mass Index (BMI)

BMI will be calculated using height (in cm) and weight (in kg) according to the formula noted below.

BMI 
$$(kg/m2)$$
 = Weight  $(kg)/[Height (cm)/100]^2$ 

#### 7.8.2 Change from baseline

Change from baseline will be calculated for each post baseline visit as follows:

Change From Baseline = Post baseline result at time - Baseline result

#### 7.8.3 Duration (days) of hospitalization during the treatment phase

The duration (days) of hospitalization during the treatment phase will be calculated using the formula noted below.

Duration (days) = (Date of discharge – Date of hospitalization) + 1

Duration (days) of hospitalization during the treatment phase will only be calculated for hospitalization(s) occurring after the date of first study treatment administration and prior to the date of last study treatment administration. For subject who remain hospitalized at the time of last treatment administration, the date of last treatment will be used for the calculation.

All deaths within 91 days will be considered censored on Day 91. Conceptually, a death corresponds to an infinite length of hospitalization but censoring at any time greater than or equal to Day 91 gives the same answer as censoring at Day 91; both correspond to giving deaths the worst rank.

In the incidence where there are multiple hospitalizations for a subject, the durations from the multiple hospitalizations will be summed to provide total duration of hospitalization for the subject.

#### 8. STATISTICAL METHODS

All statistical analyses will be performed using SAS® for Windows, version 9.4 or later. All data collected during this study will be presented in subject data listings.

All the efficacy analyses presented here will be conducted using mITT and PP populations. All safety analyses will be conducted using the Safety population.

#### 8.1 Summarizing Disposition and Baseline Data

#### 8.1.1 Subject Disposition and Withdrawals

There will be a detailed accounting of all subjects who sign an informed consent to participate in this trial.

| articipate in thi | s trial. |
|-------------------|----------|

# **8.1.2 Protocol Deviations**

Protocol deviations will be identified and classified as minor or major before un-blinding according to the following categories:

| 8.1.3 Demographics and Baseline Characteristics |
|---|
| 8.1.4 Medical History |
| Medical history will be coded using the most current available version of Medical |
| Dictionary for Regulatory Activities (MedDRA) and will be summarized by system orga |
| class (SOC) and preferred term (PT). |
| class (See e) and preferred term (1-1). |
| 8.1.5 Prior and Concomitant Medications |
| Prior medication is defined as any medication with an end date prior to the first treatment |
| date. |

| 8.1.6 Extent of Exposure and Treatment Compliance |
|---|
| 8.2 Analysis of Efficacy Data |
| The primary analysis will be conducted on the mITT population. |
| The statistical tests for the primary efficacy endpoint and secondary endpoints will be |
| two-sided with $\alpha$ =0.05. |
| 8.2.1 Primary Outcome Measure and Estimand |
| 8.2.1.1 Primary Outcome Measure |
| The primary efficacy outcome measure for this study is the change from baseline to week |
| 13 in PROMIS® Fatigue Score (T-Score). |

The Fatigue - Short Form 7a includes 7 questions and each question has a 5-point severity scale (Never, Rarely, Sometimes, Often, Always). The total score (range from 7-35) will be calculated and converted to the PROMIS® Fatigue Score (T-Score) per PROMIS

Fatigue Scoring Manual as which is included here as APPENDIX 3, Section 11.1. The higher in PROMIS® Fatigue Score (T-Score) represents the worsening of fatigue.



# 8.2.1.2 Estimand

The estimand for the primary outcome measure is described by the following attributes:

Treatment: Ampligen® vs. Placebo

**Study Population:** Adult patients with the Post-COVID Condition of fatigue.

**Primary Efficacy Variable:** Change from baseline to week 13 in PROMIS® Fatigue Score (T-Score)

**Primary Efficacy Analysis Population:** The Modified Intent-to-Treat (mITT) population is defined as the set of subjects who have received at least one dose of study treatment (Ampligen® or placebo).





#### **8.2.2** Secondary Outcome Measures

#### 8.2.2.1 Change from baseline to week 6 in PROMIS® Fatigue Score (T-Score)

Note: Additional PROMIS® Fatigue Score analysis (change from baseline) at week 6 and 13 will be performed excluding response to item, "How often did you have enough energy to exercise strenuously?"

Similar analysis methods used for the primary endpoint will be applied to analyze the data from this outcome measure.

# 8.2.2.2 Change from baseline to week 6 and 13 in distance traveled during a 6-minute walk test

The 6-minute walk test (6MWT) will be assessed throughout the study. The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

Similar analysis methods used for the primary endpoint will be applied to analyze the data from this outcome measure.

8.2.2.3 <u>Proportion of subjects with minimal clinically important difference (MCID),</u> defined as at least 54 m, in the Six-Minute Walk Test (6MWT) at the end of 12-week <u>treatment phase</u>

# 8.2.2.4 <u>Change from baseline to week 6 and 13 in PROMIS® Cognitive Function Score</u> (T-Score)

The Cognitive Function - Abilities - Short Form 8a includes 8 questions and each question has a 5-point severity scale from not at all to very much (1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, and 5=Very much) ranged from 8-40. PROMIS® Cognitive Function Score (T-Score) will be converted from the total Short Form 8a score per PROMIS Fatigue Scoring Manual which is included here as APPENDIX 3, Section 11.2. The higher in PROMIS® Cognitive Function Score (T-Score) represents the better cognitive function.

Similar

analysis methods used for the primary endpoint will be applied to analyze the data from this outcome measure.

# 8.2.2.5 <u>Change from baseline to week 6 and 13 in PROMIS® Sleep Disturbance Score</u> (T-Score)

The Sleep Disturbance - Short Form 4a includes 4 questions with three 5-point severity scales from not at all to very much (1 or 5=Not at all, 2 or 4=A little bit, 3=Somewhat, 4 or 2=Quite a bit, and 5 or 1=Very much) and very poor to very good (5=Very poor, 4=Poor, 3=Fair, 2=Good, and 1=Very good) ranged from 4-20. PROMIS® Sleep Disturbance Score (T-Score) will be converted from the total Short Form 4a score per PROMIS Fatigue Scoring Manual which is included here as APPENDIX 3, Section 11.3. The higher in

| PROMIS® Sleep Disturbance Score (T-Score) represents the worsening of sleep |
|---|
| disturbance. |
| Similar |
| analysis methods used for the primary endpoint will be applied to analyze the data from |
| this outcome measure. |
| 8.2.3 Exploratory Outcome Measures |
| 8.2.3.1 Change from baseline in COVID-19-related symptoms using Symptom Burden |
| Questionnaire for Long COVID (SBQ-LC) during the course of the treatment phase |
| Similar analysis methods used for the primary endpoint will be applied to analyze the data |
| from this outcome measure. |
| 8.2.3.2 Change from baseline in cognitive function as measured by Montreal Cognitive |
| Assessment (MoCA) at week 4, 8, and 13 during the treatment phase |
| Similar analysis |
| methods used for the primary endpoint will be applied to analyze the data from this |
| outcome measure. |
| outcome measure. |
| 8.2.3.3 <u>Incidence of hospitalization during the treatment phase</u> |
| The proportion of subjects with at least one hospitalization during the treatment phase will |
| be presented for the two treatment groups. |

# 8.2.3.4 <u>Duration (days) of hospitalization during the treatment phase</u>

| The duration (days) of hospitalization during the treatment phase will be calculated using the formula stated in Section 7.8.4. |
|---|
| the formula stated in Section 7.8.4. |
| 8.2.3.5 Evaluation of lymphocyte profile by flow cytometry in patients with post-COVID- |
| 19 conditions |
| Similar |
| analysis methods used for the primary endpoint will be applied to analyze the data from<br>this outcome measure. |
| 8.2.3.6 <u>Identification and evaluation of plasma protein biomarkers in patients with post-COVID-19 conditions</u> |

# 8.3 Analysis of Safety Data

All safety analyses will be conducted using the Safety population. All data collected will be summarized according to the variable type. No inferential statistics are planned.

| 8.3.1 Adverse Events | |
|---|---|
| Adverse events will be classified by system organ class (SOC) and preferred term (P according to the most recent version of MedDRA dictionary. | Τ) |
| TEAE are defined as adverse events with onset date on or after the first treatment. TEAE | Es |
| will be summarized by treatment group, System Organ Class, and preferred term. T | he |
| following TEAE summaries will be provided: | |
| a) Overall (i.e., regardless of severity or relationship to treatment) | |
| b) Adverse events by severity | |
| c) Related adverse events by severity | |
| d) Adverse events leading to treatment discontinuation by severity | |
| e) Adverse events leading to death by severity | |
| 8.3.2 Clinical Laboratory Evaluations | |
| 8.3.2.1 <u>Laboratory Values over Time</u> | |
| as appropriate for the variable type. | ed |
| 8.3.2.2 <u>Individual Patient Changes</u> | |

# 8.3.2.3 <u>Individual Abnormalities</u>

| 8.3.3 Vital Signs |
|---|
| Vital sign assessments are performed in order to characterize basic body function. The |
| parameters collected in this study are: systolic BP (mmHg), diastolic BP (mmHg), |
| temperature ( <sup>0</sup> C), heart rate (bpm), respiratory rate (bpm). |
| 8.3.3.1 <u>Vital Signs Values over Time</u> |
| 8.3.3.2 <u>Individual Patient Changes on Notable Vital Sign Values</u> |
| Clinically notable elevated values |
| Clinically notable below normal values |

| The EC | Electrocardiogram (ECGs) CG parameters include ventricular rate al (msec), QT interval (msec), and QTc | (beats per minute), PR interval (msec), QRS interval (msec). |
|---|---|---|
| 8.3.4.1 | ECG Values over Time | |
| 8.3.4.2 | 2 Individual Patient Changes on Notab | ole ECG Values |

| 8.3.4.3 <u>Individual Patient Changes on Interpretation</u> | |
|-------------------------------------------------------------|---|
| 8.3.5 Pulse Oxygen Saturation (SpO2) | |
| 8.3.6 Physical Examination | |
| 8.3.7 Urine Pregnancy Test | l |
| 8.3.9 SARS-CoV-2 (COVID-19) Qualitative Test | |

| 8.3.10 | <b>COVID-19 History</b> |
|--------|-------------------------|

# 9. APPENDIX 1

FIGURE 9-11: SCHEDULE OF ASSESSMENTS V1 TO V14

| Procedure/Assessments | Screening Visit | Treatment Visits | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 |
| Week | Week 0 | 1(Day 0) | 1 | 2 | 2 | 3 | 3 | 4 | 4 | 5 | 5 | 6 | 6 | 7 |
| Window Period | | Within 7<br>days of<br>SV | | | | | | . • | 192 | | | | | 7 |
| | X | | | | | | | | | | | | | |
| | X | X | | | | | | , | | | | | | |
| | X | | | | | | | | | | | | | |
| | X | X | | | | | | a. | | | | (E) (E) | | |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | | | | | | 7 | | | | X | | |
| | X | X | | | | | | | | | | X | | |
| | X | X | | X | | X | | X | | X | | X | | X |
| _ | | X | | X | | X | | X | | X | | X | | X |
| | | X | | X | | X | | X | | X | | X | | X |
| | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | X | X | - | X | | X | | X | | X | | X | |
| | X | X | | X | | X | | X | | X | | X | | X |
| | | X | | | | | | X | | | | | | |
| | X | 9 | | | | X | | | | | | X | | |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | | | | | | | | | | | | | |
| | X | X | | | | 8 8 | | | | | | X | | |

| Procedure/Assessments | Screening Visit | Treatment Visits | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 |
| Week | Week 0 | 1(Day 0) | 1 | 2 | 2 | 3 | 3 | 4 | 4 | 5 | 5 | 6 | 6 | 7 |
| | X | X | | | | | | | | | | X | | |
| | X | X | | | | | | X | X | | | | | |
| | X | X | | | | | | | | | | X | | |
| | | X | | | | | | | | | | X | | |
| | | X | | | | | | | | | | | | |
| Intervention: | | | | | | | | | | | | | | |
| | | X | | | | | | | | | | | | |
| | | X | X | X | X | X | X | X | X | X | X | X | X | X |

| -00 | 94 |
|-----|-----|
| | 8 |
| 24 | 38 |
| 5.5 | 35 |
| e j | 38 |
| | 1 |
| | 100 |
| | - 1 |
| | ŝ |
| _ | |
| | Še |
| | 9 |
| _ | |



FIGURE 9-2: SCHEDULE OF ASSESSMENTS V15 TO V27

| Procedure/Assessments | | | | | Trea | tment V | isits | | | | | Follow-up 1 | Follow-up 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V15 | V16 | V17 | V18 | V19 | V20 | V21 | V22 | V23 | V24 | V25 | Visit 26 | Visit 27 |
| Week | 7 | 8 | 8 | 9 | 9 | 10 | 10 | 11 | 11 | 12 | 12 | Week 13 (3 to<br>4 days after<br>EOT) | Week 14 |
| Window Period | | | | | | | | | | | | | ± 3 days |
| | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | | ()3 | | | .15 | | | X | | | X |
| | | | | | | | | | | X | | | X |
| | | X | | X | | X | | X | | X | | X | |
| | | X | | X | | X | | X | | X | | X | |
| | | X | | X | | X | | X | | X | | X | |
| | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | | X | | X | | X | | X | | X | | |
| | | X | | X | | X | | X | | X | | X | X |
| sment | | X | | | | | | | | | | X | |
| | | | | X | | , | - | | | | | X | |
| | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | | |
| | | | | | | | | | | | | | 3 |
| | 3 9 | | | | | | est . | | | | _ = | X | X |
| | | | 0. | 53 | | | 18 | | | | | X | X |
| | | X | X | 800 | | | 100 | | | X | | | X |
| | | | | 65 | | | | | | | | X | X |

| Procedure/Assessments | | | | Follow-up 1 | Follow-up 2 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V15 | V16 | V17 | V18 | V19 | V20 | V21 | V22 | V23 | V24 | V25 | Visit 26 | Visit 27 |
| Week | 7 | 8 | 8 | 9 | 9 | 10 | 10 | 11 | 11 | 12 | 12 | Week 13 (3 to<br>4 days after<br>EOT) | Week 14 |
| Window Period | | | | | | | | | | | | | ± 3 days |
| | | | | 33 S | | | | | | | | X | |
| | | | | | | | 10 | | | | | X | |
| | 8 | | | | | | | | | | | | |
| | X | X | X | X | X | X | X | X | X | X | X | | |

| <u> </u> |
|----------|
| <u></u> |



#### 10. APPENDIX 2

10.1 Planned by-subject listings



10.2 Planned Summary Tables

# 11. APPENDIX 3

# 11.1 PROMIS FATIGUE SCORING TABLE



# 11.2 PROMIS COGNITIVE FUNCTION SCORING TABLE



# 11.3 PROMIS SLEEP DISTURBANCE SCORING TABLE



#### 12. REFERENCES

- 1. ASA Ethical Guidelines for Statistical Practice (2016)
- 2. The Royal Statistical Society: Code of Conduct (2014)
- 3. ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3, 1996)
- 4. ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3(R1), 2013)
- 5. ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9, 1998)
- 6. ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9(R1), 2017)

# 13. VERSION HISTORY

| <b>T</b> 7 • | - | ^ |
|--------------|----|---|
| Version | Ι. | U |

This is the first final version of this document.

| <u> </u> |
|----------|